CLINICAL TRIAL: NCT00980434
Title: The Clinical Use of S-100B and NSE in Spinal Cord Injuries
Brief Title: S-100B and Neuron-specific Enolase (NSE) in Spinal Trauma
Acronym: WBS
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Wolf Harald Dr., Department for Trauma Surgery
Other Study IDs: Wolf-4
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2011-07

CONDITIONS: Spinal Cord Injury
Keywords: vertebral fracture; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum probe
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: patients with neurological symptoms
- 2: patients without neurological symptoms

SUMMARY:
The investigators are studying the clinical worth of the serum markers S-100B and NSE in patients with spinal cord injuries e.g. in patients with vertebral fractures. If there is a injury to the neuronal structures these two proteins could be secreted into the serum and add evidence to the severity of the injury.

ELIGIBILITY:
Inclusion Criteria:

* vertebral fracture
* injuries to the vertebral spine

Exclusion Criteria:

* head trauma
* polytrauma

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients from daily practice
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-02; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Neurological Symptoms | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vilmos Vecsei, M.D. Professor, Study Chair — Head of Department
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Loy DN, Kim JH, Xie M, Schmidt RE, Trinkaus K, Song SK. Diffusion tensor imaging predicts hyperacute spinal cord injury severity. J Neurotrauma. 2007 Jun;24(6):979-90. doi: 10.1089/neu.2006.0253. PMID 17600514
- [Background] Marquardt G, Setzer M, Seifert V. Serum biomarkers for experimental acute spinal cord injury: rapid elevation of neuron-specific enolase and S-100 beta. Neurosurgery. 2006 Mar;58(3):E590; author reply E590. doi: 10.1227/01.NEU.0000207967.91316.8D. No abstract available. PMID 16528168
- [Background] Marquardt G, Setzer M, Seifert V. Protein S-100b for individual prediction of functional outcome in spinal epidural empyema. Spine (Phila Pa 1976). 2004 Jan 1;29(1):59-62. doi: 10.1097/01.BRS.0000103661.78939.02. PMID 14699277
- [Background] Marquardt G, Setzer M, Seifert V. Protein S-100b as serum marker for prediction of functional outcome in metastatic spinal cord compression. Acta Neurochir (Wien). 2004 May;146(5):449-52. doi: 10.1007/s00701-004-0242-3. Epub 2004 Mar 22. PMID 15118880